CLINICAL TRIAL: NCT00374959
Title: The Prevention of Primary Endogenous Ventilator-Associated Pneumonia: A Multicenter Randomized Trial Comparing Continuous Aspiration of Subglottic Content and a 3-Day Course of Ceftriaxone.
Brief Title: Prevention of Pneumonia Comparing Ceftriaxone With Subglottic Aspiration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Principe de Asturias (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TABASCO
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2006-09-26 (Estimated); Status verified 2006-09

CONDITIONS: Pneumonia
Keywords: Prevention of pneumonia; ceftriaxone; continuous aspiration; subglottic secretions; Mechanical ventilation with Endotracheal intubation.; Absence of infection
MeSH Terms: conditions — Pneumonia | interventions — Ceftriaxone

INTERVENTIONS:
Drug: ceftriaxone
Device: Endotracheal tube for aspiration of subglottic secretions.

SUMMARY:
The primary purpose of the trial is to compare the efficacy and safety of two measures which claim to prevent early-onset ventilator-associated pneumonia.

DETAILED DESCRIPTION:
Background: In a previous double-blind, placebo-controlled, randomized trial we found that a 3-day-course of ceftriaxone significantly reduced the incidence of early-onset ventilator-associated pneumonia (EOP). Continuous aspiration of secretions accumulating in the subglottic space above the cuff of the endotracheal tube has also been shown to prevent EOP.

Objective: To compare the effect of both preventive measures on the incidence of EOP.

Design: Randomized, multicenter.

Setting: Three general intensive care units at university hospitals in Spain. Patients: Patients without signs of infection and no concomitant systemic antibiotics were included if expected to require endotracheal intubation exceeding 2 days.

Intervention: All patients were intubated with an endotracheal tube equipped with a port for aspiration of subglottic secretions and subsequently randomized to receive a three day course of 2 gram/day iv ceftriaxone without aspiration of subglottic secretions or continuous aspiration of subglottic secretions.

Measurements: All ICU-acquired infections, antibiotic therapy, colonization and infection with 3rd-generation cephalosporin-resistant microorganisms, duration of intubation and ICU-stay and-mortality.

ELIGIBILITY:
Inclusion Criteria:

* Endotracheal intubation with endotracheal tube equipped with port for aspirations of subglottic contents and expected to exceed 48 hors.
* Absence of infection.
* 18 years or older.
* Informed Consent.

Exclusion Criteria:

* Endotracheal intubation prior to admission to hospital.
* Allergic to beta-lactam antibiotics.
* Formal indication for systemic antibiotic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2000-10; Study Completion 2003-10

PRIMARY OUTCOMES:
Cumulative incidence of early-onset ventilator-associated pneumonia

SECONDARY OUTCOMES:
All ICU-acquired infections.
Duration of antibiotic therapy.
Third-generation cephalosporin resistance.
Duration of intubation and ICU-stay.
ICU-Mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Sanchez, MD, PhD, Principal Investigator — Hospital Universitario Principe de Asturias
Locations (3):
- Spain (3):
  - Francisco Alvarez Lerma, Barcelona, Barcelona
  - Miguel Sanchez Garcia, Alcalá de Henares, Madrid
  - Enrique Cerda Cerda, Getafe, Madrid

REFERENCES:
- [Background] van Saene HK, Damjanovic V, Murray AE, de la Cal MA. How to classify infections in intensive care units--the carrier state, a criterion whose time has come? J Hosp Infect. 1996 May;33(1):1-12. doi: 10.1016/s0195-6701(96)90025-0. No abstract available. PMID 8738198
- [Background] Sanchez Garcia M, Cambronero Galache JA, Lopez Diaz J, Cerda Cerda E, Rubio Blasco J, Gomez Aguinaga MA, Nunez Reiz A, Rogero Marin S, Onoro Canaveral JJ, Sacristan del Castillo JA. Effectiveness and cost of selective decontamination of the digestive tract in critically ill intubated patients. A randomized, double-blind, placebo-controlled, multicenter trial. Am J Respir Crit Care Med. 1998 Sep;158(3):908-16. doi: 10.1164/ajrccm.158.3.9712079. PMID 9731025
- [Background] Valles J, Artigas A, Rello J, Bonsoms N, Fontanals D, Blanch L, Fernandez R, Baigorri F, Mestre J. Continuous aspiration of subglottic secretions in preventing ventilator-associated pneumonia. Ann Intern Med. 1995 Feb 1;122(3):179-86. doi: 10.7326/0003-4819-122-3-199502010-00004. PMID 7810935